CLINICAL TRIAL: NCT04509752
Title: Experiences in Dysphagia Management During COVID-19 Pandemic
Brief Title: Dysphagia Management During COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SELEN SEREL ARSLAN, Principal Investigator, Hacettepe University
Other Study IDs: Dysphagia during COVID-19
Record Dates: First submitted 2020-08-11; First posted 2020-08-12 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Dysphagia; Covid19
Keywords: dysphagia; COVID-19
MeSH Terms: conditions — Deglutition Disorders; COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dysphagia clinicians: Clinicians from swallowing centers (from all over the world)
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — An online survey will be sent to each clinic to answer the survey questions.

SUMMARY:
The current study is aimed to determine the procedures applied in the dysphagia clinics during the COVID-19 pandemic period. A questionnaire consisting of 30 questions will be implemented. Each participant will be asked to answer the questions.

DETAILED DESCRIPTION:
The current study is aimed to understand the current clinical conditions and current practice regarding dysphagia management during the pandemic period/normalization period. It is a cross sectional online survey study. The first part is the survey development and testing, the second part is determination of swallowing centers and last part is survey distribution by google forms. A coordinator will be selected for each center to discuss the survey with the entire team and reply the questions.

ELIGIBILITY:
Inclusion Criteria:

* Working on a dysphagia clinic from all over the world

Exclusion Criteria:

* Not willing to participate
* Not working on a dysphagia clinic

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Clinicians who work on a dysphagia clinic will be included.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Online survey | 3 months
  An online survey will be designed to understand the current clinical conditions and current practice regarding dysphagia management during the pandemic period/normalization period

CONTACTS AND LOCATIONS:
Overall Officials: SELEN SEREL ARSLAN, Principal Investigator — Hacettepe University
Locations (1):
- Hacetttepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No